CLINICAL TRIAL: NCT01746784
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study of N6022 to Evaluate Safety and Pharmacokinetics in Subjects With Cystic Fibrosis Homozygous for the F508del-CFTR Mutation (SNO1)
Brief Title: Safety and Pharmacokinetic Study of N6022 in Subjects With Cystic Fibrosis Homozygous for the F508del-CFTR Mutation
Acronym: SNO-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N6022-1CF1-04
Record Dates: First submitted 2012-12-06; First posted 2012-12-11 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; F508del-CFTR; N6022; S-Nitrosoglutathione
MeSH Terms: conditions — Cystic Fibrosis | interventions — N6022; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N6022 (Experimental): Subjects randomized to study drug will receive N6022 by intravenous infusion once per day for 7 days
  Interventions: Drug: N6022
- Normal saline (Placebo Comparator): Subjects randomized to placebo will receive normal saline administered intravenously using the same volume as the active drug group
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: N6022 — Intravenous solution of N6022 in normal saline administered by infusion pump over 1-8 minutes depending on the dose
  Other Names: GSNORi
  Arms: N6022
Drug: Normal saline — Intravenous solution of 0.9% (weight/volume) NaCl administered by infusion pump over 1-8 minutes depending on dose of active drug used in same cohort
  Other Names: Placebo
  Arms: Normal saline

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of N6022, and to obtain descriptive information on the effect of N6022 on biomarkers of CFTR function and inflammation in adult cystic fibrosis subjects who are homozygous for the F508del-CFTR mutation.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, multicenter, sequential dose-escalation study which will occur in two parts. All selection criteria, assessments and procedures described in this protocol will be applied to both parts. Up to 5 cohorts will be studied with a total of 67 patients at approximately 18 clinical sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for F508del-CFTR gene
* Sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis
* Body weight ≥ 40 kg
* FEV1 ≥ 40% predicted
* Oxygen saturation ≥ 90% breathing ambient air
* Hematology and clinical chemistry of blood and urine results with no clinically significant abnormalities that would interfere with the study assessments
* Negative pregnancy test for women of child bearing potential
* Sexually active subjects of child bearing potential willing to follow contraception requirements

Exclusion Criteria:

* Previous enrollment in another cohort for this study.
* Any acute infection, including acute upper or lower respiratory infections and pulmonary exacerbations that require treatment within 4 weeks of Study Day 1.
* Any change in chronic therapies for CF lung disease within 4 weeks of Study Day 1.
* Blood hemoglobin <10 g/dL at screening.
* Serum albumin <2.5 g/dL at screening.
* Abnormal liver function defined as ≥ 3 x upper limit of normal (ULN) in three or more of the following: AST, ALT, GGT, ALP, total bilirubin at screening.
* History of abnormal renal function (creatinine clearance < 50 mL/min using Cockcroft-Gault equation) within a year at screening.
* History, including the screening assessment, of ventricular tachycardia or other ventricular arrhythmias.
* History, including the screening assessment, of prolonged QT and/or QTcF interval (> 450 msec).
* History of solid organ or hematological transplantation.
* Intranasal medication changes within 14 days prior to Study Day 1
* Required Use of continuous (24 hr/d) or nocturnal supplemental oxygen.
* Concomitant use of any inhibitors or inducers of CYP3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Donaldson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (17):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital - Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- See also: Home page of Sponsor — http://www.n30pharma.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 Clinical Investigator Sites enrolled 66 subjects. The first patient was screened on March 5, 2013 and the last patient was seen on April 10, 2014.
Pre-assignment Details: There were 4 ascending dose cohorts starting at 5 mg and continuing with 10 mg, 20 mg and 40 mg. There was a fifth confirmatory cohort at the maximum tested dose, 40 mg. In Cohorts 1-4 approximately 9 subjects received N6022 and 3 received placebo. In the fifth cohort 11 subjects received N6022 and 7 subjects receive placebo
Groups:
- Placebo/Saline: 0.9% (weight/volume) NaCl was administered intravenously using the same volume as the active drug group.
- 5 mg/N6022; 10 mg/N6022; 20mg/N6022; 40 mg/N6022: N6022 was administered by intravenous infusion once per day for 7 days
Period: Overall Study
Arm/Group | Placebo/Saline | 5 mg/N6022 | 10 mg/N6022 | 20mg/N6022 | 40 mg/N6022
Started | 19 | 10 | 9 | 9 | 19
Enrolled | 19 | 10 | 9 | 9 | 19
Completed | 19 | 10 | 9 | 9 | 19
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Saline: Normal saline: IV solution of 0.9% (weight/volume) NaCl administered by infusion pump over 1-8 minutes
- 5mg/N6022; 10mg/N6022; 20mg/N6022; 40mg/N6022: N6022: Intravenous solution of N6022 in normal saline administered by infusion pump over 1-8 minutes once per day for 7 days
- Total: Total of all reporting groups
Arm/Group | Normal Saline | 5mg/N6022 | 10mg/N6022 | 20mg/N6022 | 40mg/N6022 | Total
Number analyzed (Participants) | 19 | 10 | 9 | 9 | 19 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (7.27) | 26.9 (6.33) | 32.3 (7.84) | 28.6 (10.3) | 28.4 (8.46) | 28.9 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 6 | 7 | 11 | 40
  Male | 9 | 4 | 3 | 2 | 8 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 10 | 9 | 9 | 19 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 19 | 10 | 9 | 9 | 19 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 10 | 9 | 9 | 19 | 66
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/^m2] — kilograms per meter square
  kg/^m2 | 21.4 (3.25) | 21.7 (4.59) | 21.7 (2.27) | 21.0 (3.80) | 22.5 (2.62) | 21.9 (3.25)
Weight [Mean (Standard Deviation); unit: kg] — kilograms
  kg | 62.9 (11.50) | 61.8 (11.73) | 59.1 (9.06) | 56.3 (13.59) | 63.8 (12.53) | 61.0 (11.96)
FEV1 (L) [Mean (Standard Deviation); unit: L] — Liter of air
  L | 2.7 (0.85) | 2.6 (0.88) | 2.2 (0.91) | 2.1 (0.66) | 2.8 (1.12) | 2.5 (0.97)
FEV1 Percent Predicted [Mean (Standard Deviation); unit: percent] — Percent Predicted FEV1 at baseline
  percent | 72.5 (23.7) | 70.7 (19.5) | 63.3 (17.5) | 63.2 (21.1) | 73.9 (21.9) | 70.1 (21.3)
Sweat Chloride [Mean (Standard Deviation); unit: mEq/L] | 100.4 (12.9) | 103.3 (6.9) | 107.3 (6.7) | 93.1 (9.2) | 100.3 (8.3) | 100.8 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Assessments are based on numbers of subjects with abnormal clinical evaluations, abnormal laboratory assessments, and adverse events.
Time Frame: Over 7 treatment days and 7 days of follow-up
Population: Treatment emergent adverse events by Grade 1 (mild) to 5 (fatal)
Measure: Number; unit: participants
Groups:
- Normal Saline: Normal saline: Intravenous solution of 0.9% (weight/volume) NaCl administered by infusion pump over 1-8 minutes
Arm/Group | Normal Saline | 5mg/N6022 | 10mg/N6022 | 20mg/N6022 | 40mg/N6022
Number analyzed (Participants) | 19 | 10 | 9 | 9 | 19
participants
  Grade 1 (mild) | 11 | 4 | 6 | 4 | 12
  Grade 2 (moderate) | 6 | 3 | 3 | 5 | 2
  Grade 3 (severe) | 1 | 2 | 0 | 0 | 1
  Grade 4 (life threatening) | 0 | 0 | 0 | 0 | 0
  Grade 5 (fatal) | 0 | 0 | 0 | 0 | 0
  Serious TEAE | 1 | 2 | 0 | 0 | 1

2. Secondary Outcome: Change in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson standards were used to calculate percent predicted FEV1 (for age, sex, and height).
Time Frame: Change from baseline at Day 7
Population: Change in Forced Expiratory Volume in 1 second (FEV1) from baseline to Study Day 7
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- 5mg/N6022; 10mg/N6022; 20mg/N6022; 40mg/N6022: Intravenous solution of N6022 in normal saline administered by infusion pump over 1-8 minutes once per day for 7 days
Arm/Group | Normal Saline | 5mg/N6022 | 10mg/N6022 | 20mg/N6022 | 40mg/N6022
Number analyzed (Participants) | 19 | 10 | 9 | 9 | 19
percentage | 1.5 (3.44) | -0.5 (4.72) | -0.2 (3.99) | -0.7 (4.08) | 0.5 (3.04)

3. Secondary Outcome: Change in Biomarkers of CFTR Function
Description: Sweat chloride millequivalents/Liter (mEq/L)
Time Frame: Change from baseline at Day 7
Population: Change from baseline sweat chloride (mEq/L) to Study Day 14
Measure: Mean (Standard Deviation); unit: mEq/L
Groups:
- Normal Saline: Placebo will receive IV normal saline Normal saline: Intravenous solution of 0.9% (weight/volume) NaCl
- 5mg/N6022; 10mg/N6022; 20mg/N6022: N6022 by IV infusion once per day for 7 days
  N6022: Intravenous solution of N6022 in normal saline
- 40mg/N6022: N6022 by IV infusion once per day for 7 days
  N6022 in normal saline administered by infusion pump over 1-8 minutes
Arm/Group | Normal Saline | 5mg/N6022 | 10mg/N6022 | 20mg/N6022 | 40mg/N6022
Number analyzed (Participants) | 19 | 10 | 9 | 9 | 19
mEq/L | -0.2 (8.55) | -2.3 (8.12) | -2.9 (8.84) | -0.1 (11.25) | 2.9 (8.88)

ADVERSE EVENTS:
Time Frame: Through Study Day 14
Description: Adverse effect must have been present at Day 14
Arm/Group | Placebo/Saline | 5 mg/N6022 | 10 mg/N6022 | 20mg/N6022 | 40 mg/N6022
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/10 | 0/9 | 0/9 | 1/19
Other Adverse Events (participants affected / at risk) | 18/19 | 9/10 | 9/9 | 9/9 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Saline (N=19) | 5 mg/N6022 (N=10) | 10 mg/N6022 (N=9) | 20mg/N6022 (N=9) | 40 mg/N6022 (N=19)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Exacerbation of CF (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Saline (N=19) | 5 mg/N6022 (N=10) | 10 mg/N6022 (N=9) | 20mg/N6022 (N=9) | 40 mg/N6022 (N=19)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Parosmia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Chest tightness (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Infective Pulmonary Exacerbations of CF (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days